CLINICAL TRIAL: NCT03943316
Title: Single Institution (UNM) Prospective Laboratory Study of Cancer and Immune Cells in the Ascites Fluid of Ovarian Cancer Patients to Test Alternative Therapies
Brief Title: Laboratory Study of Cancer & Immune Cells in Ascites Fluid of Ovarian Cancer Patients to Test Alternative Therapies
Status: Recruiting | Type: Observational
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST UNM 1509
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Ascites
MeSH Terms: conditions — Ovarian Neoplasms; Ascites

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ascites fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ascites samples from women undergoing surgery for ovarian cancer will be collected for use in translational research.

DETAILED DESCRIPTION:
The purpose of this study is to collect ascites fluid obtained from ovarian cancer patients during cytoreductive surgery or paracentesis at the University of New Mexico Hospital or Cancer Center. Cancer cells and immune cells from the ascites fluid will be used to test novel immunotherapies for ovarian cancer treatment and to establish patient derived xenograft models to perform preclinical testing on a cancer cell population that better models the heterogeneity in patient disease

ELIGIBILITY:
Inclusion Criteria:

* All female participants, regardless of ethnicity, who are undergoing cytoreductive surgery for ovarian cancer are eligible for this study
* All participants will be eighteen years old or older
* Patients must be suspected of having a pathological diagnosis or clinical suspicion of ovarian cancer and be scheduled for surgery for tumor resection.
* Ability to understand and the willingness to sign a written informed consent document.
* Pathologic confirmation of a diagnosis of epithelial adenocarcinoma of the ovary, fallopian tube, or primary peritoneal cancer (serous, mucinous, clear cell, endometrioid, undifferentiated, mixed, transitional cell)
* Women of childbearing potential must have a negative qualitative serum pregnancy test ≤ 2 weeks prior to study entry.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

* We do not intend to include participants if they are unable to provide informed consent for this study themselves (e.g. mentally ill patients who require health care proxies to consent for any medical intervention), or vulnerable populations such as prisoners.
* Minors under age eighteen.
* Pregnant women.
* Final pathologic diagnosis that does not confirm invasive epithelial ovarian, tubal, or primary peritoneal cancer

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All female participants, regardless of ethnicity, who are undergoing cytoreductive surgery for ovarian cancer are eligible for this study; All participants will be eighteen years old or older; Patients must be suspected of having a pathological diagnosis or clinical suspicion of ovarian cancer and be scheduled for surgery for tumor resection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-12-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Collect ascites fluid obtained from ovarian cancer patients during cytoreductive surgery or paracentesis | 5 years
  To elucidate the conditions of the tumor environment that contribute to cancer dissemination in the peritoneal cavity through ex vivo evaluation of malignant ascites collected from women with ovarian, tubal, or primary peritoneal cancer.

SECONDARY OUTCOMES:
To correlate specific features of peritoneal cell populations or soluble factors with patient outcome. | 5 years
  To correlate specific features of peritoneal cell populations or soluble factors with patient outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Adams, MD, Principal Investigator — UNM Comprehensive Cancer Center
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No